CLINICAL TRIAL: NCT03654612
Title: A Single Arm,Open Clinical Study of Apatinib Combined With S-1 for the Treatment of Recurrent/Metastatic Head and Neck Malignancies
Brief Title: Apatinib Combined With S-1 for the Treatment of Recurrent/Metastatic Head and Neck Malignancies
Acronym: Y-HR2017-025
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: China International Medical Foundation (Other)
Collaborators: Chinese Society of Clinical Oncology (Other)
Responsible Party: Principal Investigator, Ping Liu, Attending doctor in oncology, China International Medical Foundation
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ChinaIMF-LP02
Record Dates: First submitted 2018-08-27; First posted 2018-08-31 (Actual); Last update posted 2018-10-18 (Actual); Status verified 2018-10

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — apatinib; S 1 (combination)

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Apatinib+S-1 (Experimental): Patients with recurrent/metastatic head and neck malignancies received apatinib plus S-1 as second-line therapy.
  Interventions: Drug: Apatinib

INTERVENTIONS:
Drug: Apatinib — Apatinib 500mg qd plus S-1 50mg bid d1-d14/28d cycle
  Other Names: S-1

SUMMARY:
This open, single-arm, exploratory study looked at the efficacy and safety of apatinib in combination with S-1 as second-line treatment of advanced head and neck malignancies.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old, male or female;
2. Pathologically diagnosed advanced head and neck malignant tumors with measurable lesions (spiral CT scan ≥10mm, meeting RECIST 1.1 criteria);
3. Late, recurrent or metastatic malignant tumors of the head and neck that are inoperable and radiotherapy;
4. According to CTCAE 4.0 and the patient's complaint, the investigator judged patients who were intolerable by second-line combined chemotherapy;
5. ECOG PS: 0-1 points;
6. Baseline blood and biochemical indicators meet the following criteria:

   Hemoglobin ≥ 80g/L, Absolute neutrophil count (ANC) ≥1.5×109/L, Platelets ≥ 90×109/L, ALT, AST ≤ 2.5 times the normal upper limit, ≤ 5 times the normal upper limit (with liver metastases), Serum total bilirubin ≤ 1.5 times the normal upper limit, Serum creatinine ≤ 1.5 times the normal upper limit, Serum albumin ≥ 30g / L;
7. The expected survival period is ≥3 months;
8. Women of childbearing age must undergo a pregnancy test (serum or urine) within 7 days prior to enrollment and the results are negative, and are willing to use appropriate methods of contraception during the trial and 8 weeks after the last administration of the test drug. For men, surgery should be sterilized, or consent should be used during the trial and 8 weeks after the last administration of the test drug.
9. Subjects volunteered to participate in the study, signed informed consent, and were well-adhered to follow-up.

Exclusion Criteria:

1. A person who has been confirmed to be allergic to apatinib and/or its excipients;
2. Patients with hypertension and antihypertensive medication can not be reduced to normal range (systolic blood pressure >140 mmHg, diastolic blood pressure >90 mmHg), with grade I or higher coronary heart disease, grade I arrhythmia (including QTc interval prolongation) Male > 450 ms, female > 470 ms) and grade I cardiac insufficiency; urine protein positive patients;
3. Have multiple factors affecting oral medications (such as inability to swallow, nausea, vomiting, chronic diarrhea, and intestinal obstruction);
4. Patients who have used apatinib or tigeo in the first line
5. abnormal blood coagulation (INR>1.5, APTT>1.5 ULN), with bleeding tendency;
6. Patients with central nervous system metastases;
7. Pregnant or lactating women;
8. Patients with other malignancies within 5 years;
9. Patients with a history of psychotropic substance abuse who are unable to quit or have a mental disorder;
10. Patients who have participated in other drug clinical trials within 4 weeks;
11. Have received VEGFR inhibitors such as sorafenib and sunitinib;
12. According to the investigator's judgment, there are serious patients who are at risk to the patient's safety or affect the patient's accompanying disease to complete the study;
13. The investigator believes that it is not suitable for inclusion.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-10-16 (Actual); Primary Completion 2020-03-01 (Estimated); Study Completion 2021-09-01 (Estimated)

PRIMARY OUTCOMES:
PFS | 40 months
  Progression free survival

SECONDARY OUTCOMES:
OS | 40 months
  Overall survival

CONTACTS AND LOCATIONS:
Locations (1):
- the Second Xiangya Hospital, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: Yes